CLINICAL TRIAL: NCT06165510
Title: Convergent Ablation Plus Left Atrial Appendage Isolation for the Treatment of Persistent Atrial Fibrillation
Acronym: CLIP-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: AtriCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 320553
Record Dates: First submitted 2023-08-15; First posted 2023-12-11 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Persistent Atrial Fibrillation; Atrial Fibrillation, Persistent; Atrium; Fibrillation; Atrial Arrhythmia
Keywords: Catheter ablation; Convergent procedure; Left atrial appendage; Hybrid ablation; Cardiac arrhythmias
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: Clinical study with 1:1 recruitment in each arm - Convergent AF Ablation with LARIAT procedure versus endocardial catheter ablation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Convergent AF Ablation with Left Atrial Appendage Exclusion (Experimental): Two Staged Convergent AF Ablation Procedure
  Stage 1 - Minimally Invasive Surgical Epicardial Ablation Procedure with concomitant LAA exclusion (LARIAT procedure)
  Stage 2 - Percutaneous Endocardial Catheter Ablation
  Interventions: Device: Epicardial AF ablation using AtriCure EPi-Sense-AF Guided Coagulation System with Left Atrial Appendage Exclusion using the AtriCure LARIAT Suture Delivery Device.; Procedure: Standard Endocardial Catheter Ablation
- Standard Endocardial Catheter Ablation (Active Comparator): Standard Endocardial Catheter Ablation
  Interventions: Procedure: Standard Endocardial Catheter Ablation

INTERVENTIONS:
Device: Epicardial AF ablation using AtriCure EPi-Sense-AF Guided Coagulation System with Left Atrial Appendage Exclusion using the AtriCure LARIAT Suture Delivery Device. — 2 stage procedure - minimally-invasive epicardial ablation with left atrial appendage exclusion using LARIAT procedure via a subxiphoid incision. This is then combined with endocardial radiofrequency catheter ablation in a separate staged procedure.
  Arms: Convergent AF Ablation with Left Atrial Appendage Exclusion
Procedure: Standard Endocardial Catheter Ablation — Standard percutaneous endocardial catheter ablation of atrial fibrillation

SUMMARY:
A randomised controlled clinical trial to assess efficacy of convergent ablation with the LARIAT procedure, as compared to standard endocardial catheter ablation in patients with long-standing persistent atrial fibrillation (AF).

DETAILED DESCRIPTION:
Atrial Fibrillation is the commonest arrhythmia and is a major cause of morbidity and mortality, often causative in ischaemic strokes and compounded by heart failure. Treatment options are limited for persistent long-standing AF (PeAF), with pulmonary vein isolation by endocardial ablation being insufficient and further additive endocardial lesions with repeated ablations yield mixed results resultant in further atrial arrhythmias. Currently success rates for catheter ablation are moderate at 40 to 70% in a single procedure.

If this was improved, patient quality of life and readmission rates would significantly improve as well as a reduction in anti-arrhythmic drug use.

The Convergent procedure - is a two stage minimally invasive hybrid approach. The first stage employs surgical ablation to the posterior wall of the left atrium in combination with the LARIAT procedure to isolate the left atrium appendage (LAA). The second stage involves endocardial catheter ablation to confirm the surgical ablation lesions, and perform further endocardial catheter ablation to leverage both epicardial and endocardial lesions to create durable, transmural lesions.

Patients with long-standing persistent AF will be randomised in a 1:1 ratio to either the Convergent ablation with the LARIAT procedure or the standard endocardial catheter ablation.

This feasibility study would assess recruitment to the trial, safety and efficacy of the Convergent procedure, in combination with a left atrial appendage system.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years; < 80 years
* Persistent AF > 1-year duration
* Left atrium size < 6cm
* Pts should be able to provide written informed consent.

Exclusion Criteria:

* Subjects currently enrolled in another investigational study except in case of observational registry with no associated treatments.
* Subject has a reversible cause of AF or transient AF
* Subject is absent of LAA or if the LAA is previously surgically ligated
* Subject has had previous cardiac surgery or abdominal surgery.
* Subject has contraindication to anticoagulation.
* Patients with hypertrophic cardiomyopathy.
* Patients with significant valve disease.
* Subject has had previous catheter or surgical ablation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Demonstrate trial feasibility with regards to recruitment rate | 24 months
  Recruitment rate to the Convergent Procedure (with LARIAT) and radiofrequency ablation in the cohort of patients with our specific inclusion criteria will be measured.
A composite of major adverse events (MAE) and complications occurring within 30 days post procedure will be measured. | 30 days post procedure
  Primary safety endpoint was a composite of major adverse events (MAE) and complications occurring within 30 days post procedure. Any of the following endpoints counted as a MAE: death, stroke/transient ischaemic attack, myocardial infarction, pericarditis requiring pericardiocentesis or prolongation of hospital stay or readmission, cardiac perforation/tamponade, bleeding at vascular access site requiring intervention, pneumothorax requiring intervention (after removal of chest drain, symptomatic pulmonary vein stenosis > 70%, permanent phrenic nerve paralysis, atrio-oesophageal fistula, major vascular complications and infection at surgical or puncture site requiring surgical intervention.
Success or failure at 12 months of persistent AF patients to be free of: Atrial arrhythmia (classed as documentation of atrial fibrillation, atrial flutter or atrial tachycardia lasting for more than 30 seconds) | Measured from the end of a 3 month blanking period to 12 months post procedure
  Recurrence of any atrial arrhythmia > 30 seconds on or off class I / III medications
Measure improvement in symptoms following convergent ablation | 12 months
  Measure change in quality of life through the European Heart Rhythm Association (EHRA) patient survey which categorises patients symptoms during physical activity in 4 categories. The higher the class, the greater the severity of symptoms with Class 1 indication no symptoms and Class 4 indicating disabling symptoms with discontinuation of normal daily activity.

SECONDARY OUTCOMES:
Measure improvement in symptoms following convergent ablation. | 12 months
  To measure improvement in quality of life assessment measured through the Atrial Fibrillation Effect on QualiTy-of-Life (AFEQT) questionnaire) to be performed at baseline, 6 months and 12 months post procedure. This survey employs the use of 20 questions regarding symptoms, effect on daily activities, treatment concerns and treatment satisfaction to generate a score from 0 - 100. The lower the score, the more severe the disability with score 0 indicating complete disability and score 100 indicating no disability or limitation in daily activities.
Changes in baseline left ventricular ejection fraction (LVEF) in patients with severe left ventricular systolic dysfunction (EF <35%) will be measured. | 12 months
  Assessment of LVEF via transthoracic echocardiogram at baseline and transthoracic echocardiogram at 12 months post procedure.
Measure improvement in NYHA (New York Heart Association) class in patients with NYHA class III to IV following convergent AF ablation. | 12 months
  Assessment of heart failure symptoms and functional status via clinic review at baseline and 12 months post-procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Ahsan, Principal Investigator — Consultant Cardiologist and Electrophysiologist, Barts Health NHS Trust
Locations (1):
- St Bartholomew's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No